CLINICAL TRIAL: NCT01176526
Title: The Role of Social Comparisons in Coping and Quality of Life Following a Prostate Cancer Diagnosis
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999910172; 10-HG-N172
Record Dates: First submitted 2010-08-05; First posted 2010-08-06 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2016-01-27

CONDITIONS: Prostate Cancer
Keywords: Coping; Quality of Life; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
Social comparisons may function as a coping strategy, but their role in coping and quality of life has not been well characterized. The purpose of the current study is to investigate the relationships between cognitive appraisals; coping strategies; social comparisons; and quality of life among men with prostate cancer. The conceptual framework for this study is drawn from Festinger s Social Comparison Theory, Lazarus and Folkman s Transactional Model of Stress and Coping, and Mishel s Uncertainty in Illness Theory. A cancer diagnosis is accompanied by uncertainty about how cancer will affect one s life. Theory and empirical data suggest that in conditions of uncertainty, coping affects adjustment to a condition. Social comparisons have been postulated to be more prevalent in uncertain situations. Because little is known about how social comparisons operate, participants in this study will be recruited exclusively from prostate cancer support groups. Support groups provide a context in which individuals are likely to make social comparisons and to be cognizant of these comparisons. Prostate cancer provides a model of a common, chronic condition with complex etiology. Prostate cancer treatment may cause sexual, urinary, and bowel side effects, which may affect patients quality of life and elicit attempts to cope. One way of managing the prostate cancer experience may be to compare oneself to others who are doing better or worse than oneself on relevant dimensions. The interpretation of social comparisons may positively or negatively affect one s perceived quality of life. There have been no studies among prostate cancer patients that have quantitatively measured the use of social comparisons. There is also a paucity of research in this population regarding the predictors of coping strategies and the predictors of quality of life across multiple domains. This study will use a cross-sectional, mixed methods survey to investigate relationships between cognitive appraisals, coping, and quality of life and to qualitatively explore social comparisons among men with prostate cancer. Participants may complete the survey on paper or online. The primary outcomes are the use of coping strategies, including social comparisons, and quality of life. Individuals with a personal or family history of prostate cancer are currently seen by genetic counselors as part of research studies investigating the genetic basis of prostate cancer. If relationships are demonstrated between the social comparisons and quality of life, genetic counselors may want to assess patients social comparisons to evaluate how patients are coping with their condition.

DETAILED DESCRIPTION:
Social comparisons may function as a coping strategy, but their role in coping and quality of life has not been well characterized. The purpose of the current study is to investigate the relationships between cognitive appraisals; coping strategies; social comparisons; and quality of life among men with prostate cancer. The conceptual framework for this study is drawn from Festinger s Social Comparison Theory, Lazarus and Folkman s Transactional Model of Stress and Coping, and Mishel s Uncertainty in Illness Theory. A cancer diagnosis is accompanied by uncertainty about how cancer will affect one s life. Theory and empirical data suggest that in conditions of uncertainty, coping affects adjustment to a condition. Social comparisons have been postulated to be more prevalent in uncertain situations. Because little is known about how social comparisons operate, participants in this study will be recruited exclusively from prostate cancer support groups. Support groups provide a context in which individuals are likely to make social comparisons and to be cognizant of these comparisons. Prostate cancer provides a model of a common, chronic condition with complex etiology. Prostate cancer treatment may cause sexual, urinary, and bowel side effects, which may affect patients quality of life and elicit attempts to cope. One way of managing the prostate cancer experience may be to compare oneself to others who are doing better or worse than oneself on relevant dimensions. The interpretation of social comparisons may positively or negatively affect one s perceived quality of life. There have been no studies among prostate cancer patients that have quantitatively measured the use of social comparisons. There is also a paucity of research in this population regarding the predictors of coping strategies and the predictors of quality of life across multiple domains. This study will use a cross-sectional, mixed methods survey to investigate relationships between cognitive appraisals, coping, and quality of life and to qualitatively explore social comparisons among men with prostate cancer. Participants may complete the survey on paper or online. The primary outcomes are the use of coping strategies, including social comparisons, and quality of life. Individuals with a personal or family history of prostate cancer are currently seen by genetic counselors as part of research studies investigating the genetic basis of prostate cancer. If relationships are demonstrated between the social comparisons and quality of life, genetic counselors may want to assess patients social comparisons to evaluate how patients are coping with their condition.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Under 70 years old (the mean age of diagnosis for prostate cancer)
* Diagnosed between ages 18 and 70 with localized prostate cancer of stage T1b, T1c, or T2

EXCLUSION CRITERIA:

- History of another primary cancer other than a skin cancer that was not melanoma

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2010-07-19; Study Completion 2016-01-27

PRIMARY OUTCOMES:
Perceived Quality of Life

SECONDARY OUTCOMES:
Use of various coping strategies
Use of Social ComparisonsUse of Various Coping Strategies

CONTACTS AND LOCATIONS:
Overall Officials: Barbara B Biesecker, Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Human Genome Research Institute (NHGRI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ahmad MM. Psychometric evaluation of the Cognitive Appraisal of Health Scale with patients with prostate cancer. J Adv Nurs. 2005 Jan;49(1):78-86. doi: 10.1111/j.1365-2648.2004.03266.x. PMID 15610384
- [Background] Bellizzi KM, Blank TO, Oakes CE. Social comparison processes in autobiographies of adult cancer survivors. J Health Psychol. 2006 Sep;11(5):777-86. doi: 10.1177/1359105306066637. PMID 16908472
- [Background] Boehmer S, Luszczynska A, Schwarzer R. Coping and quality of life after tumor surgery: personal and social resources promote different domains of quality of life. Anxiety Stress Coping. 2007 Mar;20(1):61-75. doi: 10.1080/10615800701195439. PMID 17999215